CLINICAL TRIAL: NCT02988310
Title: Comparison of Gait Characteristics in Individuals With Trans Femaoral and Trans Tibial Limb Loss
Brief Title: Comparison of Gait Characteristics in Individuals With Above and Below Knee Limb Loss
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, hhotaman, Research Assistant, PhD,PT, Hacettepe University
Other Study IDs: G10
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Amputation
Keywords: Limb Loss; Gait Characteristics

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Individuals with below knee limb loss: Individuals with below knee limb loss will be participants of the group.
  Interventions: Other: No intervention
- Individuals with above knee limb loss: Individuals with above knee limb loss will be participants of the group.
  Interventions: Other: No intervention
- Healthy individuals: Healthy individuals will be participants of the group.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Twelve individuals with above knee limb loss, 12 individuals with below knee limb loss,15 healthy individuals will be participants of the study. Participants with lower limb loss will evaluate with the following assessment tools: Demographic datas; age, gender, height, body mass will be recorded. Gait parameters (step length, variation of step length, time on each foot, ambulation index) will evaluate with Gait Trainer Biodex 2, at participant's preferred speed.

DETAILED DESCRIPTION:
Twelve individuals with above knee limb loss, 12 individuals with below knee limb loss,15 healthy individuals who were referred to receive amputee rehabilitation at Hacettepe University, Faculty of Health Sciences, department of Physiotherapy and Rehabilitation, Prosthetics and Biomechanics unit, and healthy individuals will be the subjects of this study.

Participants will evaluate with the following assessment tools: Demographic datas; age, gender, height, body mass will be recorded. Gait parameters (step length, variation of step length, time on each foot, ambulation index, gait speed) will evaluate with Gait Trainer Biodex 2, at participant's preferred speed. To eliminate the learning effect, participants practiced at treadmill to determine appropriate gait speed. Once participants implied the preferred speed, they asked to walk at their self selected speed for 6 minutes. Data was recorded between the 4nd and 6th minutes at walk.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with unilateral above knee lower limb loss and below knee limb loss
* Age between 20-55 years
* Using conventional type socket design Dynamic foot using

Exclusion Criteria:

* Have passive joint limitation at extremities
* Surgery at last 1 year
* Systemic problems such as neurological disorders, rheumatoid disorders
* Another orthopedic anomalies

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals with unilateral below or above knee limb loss
Sampling Method: Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Step length assesment while walking. | Initially evaluation at first minute

SECONDARY OUTCOMES:
Ambulation index assessment while walking. | Initially evaluation at first minute